CLINICAL TRIAL: NCT02943356
Title: Observational Study to Evaluate the Effect of Tadalafil 5mg Once Daily on Erectile Dysfunction and QOL in Andropause Patients With Erectile Dysfunction
Brief Title: Effect of Tadalafil on Erectile Dysfunction Treatment and QOL Improvement Effect (by SF-12) in Andropause Patients With Erectile Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Keun-Sang Yum, Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TEDQOL
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Erectile Dysfunction; Andropause
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tadalafil (Experimental): Patients will be treated with Tadalafil for 8 weeks.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Patients will be treated with Tadalafil for 8 weeks

SUMMARY:
Observational study to evaluate the effect of Tadalafil 5mg once daily on Erectile Dysfunction and QOL in Andropause patients with Erectile Dysfunction.

Patients will be observed for 8weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Above 35 years men
2. Approving ADAM questionnaire and andropause patients with symptoms under contents

   ; easily fatigue, decreased sexual desire, general weakness, decreasing memory ect.
3. Patient with Erectile Dysfunction above 6 months
4. International Index of Erectile Function(IIEF-5) score under 21
5. Voluntarily one want to treatment with Tadalafil 5 mg daily
6. Voluntarily one agree this study and write informed consent

Exclusion Criteria:

1. Persons who have taken PDE-5 inhibitor within last one month for Erectile Dysfunction
2. Persons who taken testosterone treatment within last one month
3. Persons who be history of Myocardiac infarction
4. The history of taken organic nitrate drug
5. The history of cardiovascular disease

   * In myocardial infarction within the last 90 days was now
   * Unstable angina or angina pectoris during intercourse that occurred
   * New York Heart Association Class 2 during the last six months or more sever cardiac failure
   * Uncontrolled arrythmia, hypotension(<90/50mmHg), or uncontrolled blood pressure(>170/100mmHg)
   * Persons who have a stroke within the last six months
6. Persons who have degrative retinal disease including Pigmentary retinites
7. Formerly persons who have one eye blindness by Artery anterior ischemic optic neuropathy with or without taking PDE5 inhibitor.
8. Persons who use inhibitor or agonist drug f Hepatic cytochrome P4503A4
9. Persons who use alpha antagonist add antihypertensive drug
10. Moderate liver or kidney failure
11. Major psychiatric or personality disorder
12. Persons have phobia trial drug
13. Persons have invasive treatment of prostate gland
14. Congenital anomaly of penis
15. Galactose, Lactose, Glucose intolerance patient
16. Research coordinators who are deemed unfit

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change on SF-12 Score from baseline to week 8 | week 0 to week 8
  The comparison of change of Quality of Live at baseline and 8 week (SF-12)

SECONDARY OUTCOMES:
Change on SF-12 Score from baseline to week 4 | week 0 to week 4
  The comparison of change of Quality of Life at baseline and 4 week (SF-12)
Change on bioimpedance Analysis from baseline to week 8 | week 0 to week 8
  The comparison of change of bioimpedance Analysis at baseline and 8 week
Change on IIEF-5 Score from baseline to week 4, week 8 | week 0 to week 4, week 8
  The comparison of score at baseline, 4 week and 8 week (IIEF-5)
Change on free radical from baseline to week 4, week 8 | week 0 to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Keun-Sang Yum, M.D., PhD, Principal Investigator — Uijeongbu St. Mary's Hospital
Locations (1):
- Uijeongbu St.Mary's Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided